CLINICAL TRIAL: NCT02019810
Title: Impact of Cardiac Blood Flow on Cerebral Blood Flow in Patients With Severe Traumatic Brain Injury
Acronym: DEBITC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-003276-13
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Severe Traumatic Brain Injury With High Cerebral Pressure
MeSH Terms: interventions — Norepinephrine; Dobutamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noradrenaline alone (Active Comparator): Treatment for 30 minutes with noradrenaline alone
  Interventions: Drug: Norepinephrine
- Noradrenaline + dobutamine (Experimental): Treatment with noradrenaline and dobutamine for 30 minutes
  Interventions: Drug: Dobutamine and norepinephrine

INTERVENTIONS:
Drug: Norepinephrine
  Arms: Noradrenaline alone
Drug: Dobutamine and norepinephrine
  Arms: Noradrenaline + dobutamine

SUMMARY:
Severe traumatic brain injury with increased intracranial pressure can lead to decreased cerebral blood flow. Low cerebral blood flow is responsible for secondary lesions, leading to bad prognosis. It is not yet established whether increasing cardiac output in these patients can lead to an increase in cerebral blood flow, although there are some arguments in favor of this hypothesis. The aim of this study is to demonstrate that increasing cardiac output will improve cerebral blood flow in patients with severe traumatic injury and high cerebral pressure.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury (TBI) with pattern of oligemia (diastolic velocity < 30cm/second and/or mean velocity < 45cm/second measured with transcranial doppler or oxygen tissue pressure < 15mmHg)
* Closed traumatic brain injury
* Isolated TBI or polytraumatism
* Age between 18 and 65 years old
* Affiliated to a social security system

Exclusion Criteria:

* Instable episodes of high cerebral pressure
* Craniectomy
* High cerebral pressure without TBI
* No autoregulation
* Current hemorrhagic shock
* Chronic cardiac failure
* Chronic renal failure
* Hyperemia measured with transcranial doppler
* Short life expectancy
* Refused consent from the family
* Protected patients by the law
* Hypersensibility to one of the treatment or sulfites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Mean blood flow velocity | After one hour of treatment
  Mean blood flow velocity averaged on the two middle cerebral arteries (right and left) measured one after after the initiation of treatment. Each velocity is calculated as an average on the 10 last minutes form continuous transcranial doppler monitoring

SECONDARY OUTCOMES:
Evolution of brain oxygenation under treatment | During one hour of treatment
  Comparison of the brain tissue oxygenation curves (PbrO2) under treatment with and without dobutamine
Dobutamine doses | After one hour of treatment
  Dobutamine doses required to reach the same cerebral perfusion pressure than noradrenaline alone
Resistivity index on renal doppler | After one hour of treatment
  Measure of resistivity index on renal doppler after one hour of treatment with and without dobutamine
Pulsatility index on renal doppler | After one hour of treatment
  Measure of pulsatility index (PI) on renal doppler before and after one hour of treatment with and without dobutamine prediction of cerebral blood flow increase (patients with high initial renal PI)
Cardiac output modifications | During one hour of treatment
  Comparison of cardiac blood flow modifications under treatment for one hour with and without dobutamine

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France